CLINICAL TRIAL: NCT04042779
Title: Development of a Model-based Working Memory Training and Investigation of Its Comparative Efficacy: A Randomized, Double-blind Study on Healthy Adults
Brief Title: Development of a Model-based Working Memory Training and Investigation of Its Comparative Efficacy
Acronym: sMarT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018-01226; me19Magon
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Working Memory
Keywords: Multiple task training; Single task training; Model-based working memory training; Cognitive training; Long-term WM capacity; near transfer effects of the training; far transfer effects of the training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- model-based WM training (Active Comparator): In order to build the model-based WM training, existing tasks used to assess the different component of the Baddeley's model will be reviewed on their findings according to test-retest reliability and construct validity. For each component - phonological loop, visuospatial sketchpad, episodic buffer and central executive - the task with the highest reliability and validity will be chosen and then build the basis for the computerized training program. This procedure results in a model-based, adaptive, computerized training program for WM.
  Interventions: Other: model-based WM training
- single-task WM training (Active Comparator): The basis for the single-task training administered to the second group will be the widely used "dual-n-back training paradigm" suggested by Jaeggi et al. (2008). A complex dual n-back task including a visual and an auditory WM task will be implemented for tablet devices.
  Interventions: Other: single-task WM training
- multiple-task WM training (Active Comparator): Verbal WM tasks - particularly letter span and digit span tasks - and a visuospatial WM task are most commonly used (e.g. Dahlin et al., 2008; Klingberg et al., 2005; Westerberg et al., 2007). Therefore, a multiple-task training including these tasks will be administered to the third group.
  Interventions: Other: multiple-task WM training
- sham intervention (Sham Comparator): Active control group that as well performs a training, however not based on WM. To exclude the involvement of WM, a motor training will be administered to the control group.
  Interventions: Other: sham intervention

INTERVENTIONS:
Other: model-based WM training — model-based WM training program: four sessions a week, 45 minutes each; lasting for three weeks
  Arms: model-based WM training
Other: single-task WM training — single-task WM training program: four sessions a week, 45 minutes each; lasting for three weeks
  Arms: single-task WM training
Other: multiple-task WM training — multiple-task WM training program: four sessions a week, 45 minutes each; lasting for three weeks
  Arms: multiple-task WM training
Other: sham intervention — motor training program: four sessions a week, 45 minutes each; lasting for three weeks
  Arms: sham intervention

SUMMARY:
This study is to investigate the efficacy of model-based Working Memory (WM) training using an appropriate control condition. The interventions are a model-based, a single-task and a multiple-task training on WM in order to compare the efficacies of these different training approaches for WM. A sham intervention acts as active control group. Each intervention will be presented on a tablet device.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature

Exclusion Criteria:

* Medical history of neurological or psychiatric disorders
* Any history of substance abuse
* Color vision deficiency
* Inability to used table devices
* Montreal Cognitive Assessment < 26

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change in Rotation Span Task Score | assessment at baseline (=T2) and 3 weeks after baseline (=T3)
  First, the distractor task is judging whether a rotated letter is presented correctly, or is a mirrored image of the letter. Second, the to-be-remembered items are arrows of either short or long length and pointing in one of eight different directions. Finally, the rotation-arrow sequence is repeated from two to five times per trial. Scores are calculated by summing the number of arrows correctly recalled in the correct order.
Change in Symmetry Span Task Score | assessment at baseline (=T2) and 3 weeks after baseline (=T3)
  First, the distractor task is judging whether a displayed shape is symmetrical along its vertical axis. Second, the to-be-remembered items are locations of red squares in a 4×4 grid of potential locations. Finally, the number of symmetry-location pairs varied from two to five times per trial. Scores are calculated by summing the number of red square locations correctly recalled in the correct order.
Change in Operation Span Task Score | assessment at baseline (=T2) and 3 weeks after baseline (=T3)
  Subjects first solve a math problem, and then see a letter, and then solve another math problem, and see another letter. This math-letter sequence is repeated from three to seven times for each trial with an unpredictable length each time. After each math-letter sequence, subjects are asked to recall, in order, the preceding letters. Scores are calculated by summing the number of letters correctly recalled in the correct order.

SECONDARY OUTCOMES:
Change in Rotation Span Task Score | assessment at baseline (=T2) and 12 weeks after baseline (=T4)
  First, the distractor task is judging whether a rotated letter is presented correctly, or is a mirrored image of the letter. Second, the to-be-remembered items are arrows of either short or long length and pointing in one of eight different directions. Finally, the rotation-arrow sequence is repeated from two to five times per trial. Scores are calculated by summing the number of arrows correctly recalled in the correct order.
Change in Symmetry Span Task Score | assessment at baseline (=T2) and 12 weeks after baseline (=T4)
  First, the distractor task is judging whether a displayed shape is symmetrical along its vertical axis. Second, the to-be-remembered items are locations of red squares in a 4×4 grid of potential locations. Finally, the number of symmetry-location pairs varied from two to five times per trial. Scores are calculated by summing the number of red square locations correctly recalled in the correct order.
Change in Operation Span Task Score | assessment at baseline (=T2) and 12 weeks after baseline (=T4)
  Subjects first solve a math problem, and then see a letter, and then solve another math problem, and see another letter. This math-letter sequence is repeated from three to seven times for each trial with an unpredictable length each time. After each math-letter sequence, subjects are asked to recall, in order, the preceding letters. Scores are calculated by summing the number of letters correctly recalled in the correct order.
Change in Trail making Test A/B | assessment at baseline (=T2) and 3 weeks after baseline (=T3) and 12 weeks after baseline (=T4)
  The Trail making Test A/B consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy with the time taken to complete the test being used as the primary performance metric
Change in Rey Auditory Verbal Learning test | assessment at baseline (=T2) and 3 weeks after baseline (=T3) and 12 weeks after baseline (=T4)
  Participants are read a list of 15 words aloud by the person administering the test. The entire test takes 10-15 minutes to administer and includes five presentations of a 15 word list (list A), followed by a free recall of a second word list (list B). Finally there is a sixth recall trial of the first list (List A). Recognition is tested by asking which of 30 words wre read aloud from list A and which were not. The words are read at a rate of one word per second. The overall goal of the task is to repeat all of the words the participant can remember in any order.
Change in Rey Osterrieth Complex Figure Test | assessment at baseline (=T2) and 3 weeks after baseline (=T3) and 12 weeks after baseline (=T
  The Rey-Osterrieth complex figure test (ROCF) is a neuropsychological assessment in which examinees are asked to reproduce a complicated line drawing, first by copying it freehand (recognition), and then drawing from memory (recall). Each copy is scored for the accurate reproduction and placement of 18 specific design elements.
Change in Raven's Progressive Matrices | assessment at baseline (=T2) and 3 weeks after baseline (=T3) and 12 weeks after baseline (=T
  The Raven's Progressive Matrices is administered as a nonverbal group test. It is typically a 60-item test used in measuring abstract reasoning and regarded as a non-verbal estimate of fluid intelligence. Many patterns are presented in the form of a 6×6, 4×4, 3×3, or 2×2 matrix, giving the test its name. All of the questions on the Raven's progressives consist of visual geometric design with a missing piece. The test taker is given six to eight choices to pick from before filling in the missing piece. Scoring on the Raven's Progressive Matrices is based on two factors: How many out of 60 matrices problems the tester correctly solved and the age of the tester. For each age group, N number of correct answers corresponds to a certain percentile score.
Change in Depression Anxiety Stress Scales | assessment at baseline (=T2) and 3 weeks after baseline (=T3) and 12 weeks after baseline (=T
  The Depression Anxiety Stress Scales is made up of 42 self-report items to be completed over five to ten minutes, each reflecting a negative emotional symptom. Each of these is rated on a four-point Likert scale of frequency or severity of the participants' experiences over the last week with the intention of emphasising states over traits. These scores ranged from 0, meaning that the client believed the item "did not apply to them at all", to 3 meaning that the client considered the item to "apply to them very much, or most of the time".

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Magon, Dr. phil., Principal Investigator — Department of Neurology, University Hospital Basel
Locations (1):
- Department of Neurology, University Hospital Basel, Basel, Switzerland